CLINICAL TRIAL: NCT02909400
Title: An Exploratory, Double-blind, Randomized, Placebo-controlled, Single-center, Two-way Cross-over Study With KH176 in Patients With the Mitochondrial DNA tRNALeu(UUR) m.3243A>G Mutation and Clinical Signs of Mitochondrial Disease
Brief Title: The KHENERGY Study
Acronym: KHENERGY
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Khondrion BV (Industry)
Collaborators: Radboud University Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: KH176-201
Record Dates: First submitted 2016-09-13; First posted 2016-09-21 (Estimated); Last update posted 2018-02-23 (Actual); Status verified 2018-02

CONDITIONS: Mitochondrial Diseases; Mitochondrial Myopathies; Mitochondrial Encephalomyopathies; MELAS; MIDD
Keywords: mitochondrial; oxidative phosphorylation (oxphos); MELAS; MIDD; KH176; Proof of Concept
MeSH Terms: conditions — Mitochondrial Diseases; Mitochondrial Myopathies; Mitochondrial Encephalomyopathies; MELAS Syndrome | interventions — 6-hydroxy-2,5,7,8-tetramethylchroman-2-carboxylic acid

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Treatment A (Experimental): Oral administration of 100 mg KH176 twice daily
  Interventions: Drug: KH176
- Treatment B (Placebo Comparator): Oral administration of matching placebo twice daily
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: KH176
  Arms: Treatment A
Drug: placebo
  Arms: Treatment B

SUMMARY:
Mitochondrial Diseases are rare, progressive, multi-system, often-early fatal disorders affecting both children and adults. KH176 is a novel chemical entity currently under development for the treatment of inherited mitochondrial diseases, including MELAS (Mitochondrial Encephalomyopathy, Lactic acidosis, and Stroke-like episodes), MIDD (Maternally Inherited Diabetes and Deafness), Leigh's Disease and LHON (Leber's Hereditary Optic Neuropathy). The current Proof of Concept study aims to explore the effects of treatment with KH176 for 4 weeks on clinical signs and symptoms and biomarkers of mitochondrial disease and to evaluate the safety and pharmacokinetics of KH176 in patients with m.3242A>G related mitochondrial disease.

DETAILED DESCRIPTION:
The trial will be a double blind, randomized, placebo-controlled, single-centre, two-way cross-over trial. Twenty patients, with a confirmed mitochondrial DNA tRNALeu(UUR) m.3243A>G mutation and with clinical signs of mitochondrial disease, will be randomized over 2 groups (active or placebo first). After a screening period and a training session, each group will have 2 dosing periods of 28 days, with a washout period of at least 28 days in between. On these occasions, patients will receive 100 mg KH176 twice daily (treatment A) or a matching placebo (treatment B) twice daily for 28 days.

Clinical assessments will be performed once in a training session prior to baseline, at baseline and in week 4 post dosing during each treatment phase (A and B). Testing conditions and circumstances, with respect to timing of the assessments, hospitalization and meals, will be standardized for each assessement period. Furthermore, assessments of biomarkers for mitochondrial functioning, pharmacokinetics and specific safety assessments will be performed weekly.

ELIGIBILITY:
Inclusion Criteria:

1. Males and females aged 18 years or older at screening
2. Ability and willingness to sign the Informed Consent Form prior to screening evaluations.
3. Confirmed mitochondrial DNA tRNALeu(UUR) m.3243A>G mutation
4. Heteroplasmy level as measured in urine ≥ 20 %.
5. Body Mass Index (BMI) 18.0-30.0 kg/m2 (extremes included) at screening
6. Clinical evidence of mitochondrial disease, positive NMDAS score (including but not limited to MELAS, MIDD and mixed types). CPEO patients with signs restricted to the eye only are not considered eligible.
7. Disease appropriate physical and mental health as established by medical history, physical examination, electrocardiogram (ECG) and vital signs recording, and results of biochemistry, hematology and urinalysis testing within 3 weeks prior to the first dose as judged by the Investigator.
8. Appropriate cardiac functioning as assessed by medical history, ECG and Echo, evaluated by a cardiologist.
9. Able to comply with the study requirements, including exercise testing and swallowing study medication
10. Willingness to use adequate contraceptive methods (male and female) and negative urine pregnancy test (females) at screening and first baseline assessment.
11. Able and willing to refrain from the use of (multi)vitamins, co-enzyme Q10, Vitamine E, riboflavin, and anti-oxidant supplements (and idebenone/EPI-743), as well as any medication negatively influencing mitochondrial functioning (including but not limited to valproic acid, glitazones, statins, anti-virals, amiodarone, and NSAID's) as well as any strong Cytochrome P450 inhibitors (all 'conazoles-anti-fungals', HIV antivirals, grapefruit) and strong Cytochrome P450 inducers (a.o. carbamazepine, phenobarbital, phenytoin, rifampicine, St Johns wort, pioglitazone, troglitazone) as well as any medication known to affect cardiac repolarization (all anti-psychotics, several anti-depressants: nor/amytriptilline, fluoxetine, anti-emetics: domperidone (motilium) granisetron, ondansetron).

Exclusion Criteria:

1. Motoric abnormalities other than related to the mitochondrial disease interfering with the outcome parameters.
2. CPEO patients with clinical signs and symptoms restricted to the eye only
3. Heteroplasmy level as measured in urine < 20%
4. Poor nutritional state as judged by the investigator
5. Body Mass Index (BMI) not within 18.0-30.0 kg/m2 at screening.
6. History of cancer
7. Surgery or active illness of gastro-intestinal tract that might interfere with absorption.
8. Participation in a trial of an investigational product in the preceding 3 months prior to the first dose or during this trial.
9. Positive drug, alcohol or cotinine test at screening and/or admission (Day 1 of the first dosing period).
10. Clinically relevant abnormal laboratory, ECG recordings, cardiac echo (within 1 year prior to screening), vital signs or physical or mental findings at screening as judged by the Investigator.
11. Clinically relevant abnormal ECG or cardiac functioning as judged by a cardiologist.
12. ECG: QTc > 450 ms, abnormal T-wave
13. Symptomatic heart failure or signs of ischemic heart disease
14. Left Ventricular Ejection Fraction <45%
15. History or family history of congenital Long QT syndrome
16. Increased or decreased potassium (local laboratory normal range)
17. Inadequate contraception use, pregnancy or breast feeding (females)
18. Clinically significant presence or history of allergy as judged by the Investigator.
19. History of hypersensitivity or idiosyncrasy to any of the components of the investigational drug.
20. Within 4 weeks prior to dosing, the use of:

    * (multi)vitamins, co-enzyme Q10, Vitamine E, riboflavin, and anti-oxidant supplements (and idebenone/EPI-743),
    * as well as any medication negatively influencing mitochondrial functioning (including but not limited to valproic acid, glitazones, statins, anti-virals, amiodarone, and NSAID's)
    * as well as any strong Cytochrome P450 inhibitors (all 'conazoles-anti-fungals', HIV antivirals, grapefruit)
    * and strong Cytochrome P450 inducers (a.o. carbamazepine, phenobarbital, phenytoin, rifampicin, St Johns wort, pioglitazone, troglitazone)
    * as well as any medication known to affect cardiac repolarization (all anti-psychotics, several anti-depressants: nor/amitriptyline, fluoxetine, anti-emetics: domperidone (motilium) granisetron, ondansetron)
    * as well as any medication metabolized by Cytochrome P450 with a narrow therapeutical width. (for reference: drug interaction table of Indiana University http://medicine.iupui.edu/clinpharm/ddis/clinical-table/)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2016-09 (Actual); Primary Completion 2017-07 (Actual); Study Completion 2017-07 (Actual)

PRIMARY OUTCOMES:
Movement disorders | one month
  Rater assessed change from baseline of motoric abnormalities and movement characteristics

SECONDARY OUTCOMES:
NMDAS | one month
  Change from baseline of the Newcastle Mitochondrial Disease Activity Score
Spirometric parameters (FVC,FEV1, PEF) | one month
  Change from baseline in spirometric parameters
Spirometric parameters (MIP, MEP) | one month
  Change from baseline in spirometric parameters
Sit to Stand Test (30 seconds) | one month
  Change from baseline assessment of the maximum number of sit-standings in 30 seconds time
Handgrip Dynamometry | one month
  Change from baseline assessment of the maximum grip strenght
6-min chewing test | one month
  Change from baseline assessment in rate of mastication
6-min chewing test | one month
  Change from baseline assessment of pain and tiredness (VAS) during a 6-min chewing test
6-MWT | one month
  Change from baseline assessment of the Distance during a 6-min Walk Test
RAND-SF36 score | one month
  Change from baseline in the RAND-SF36
HAD and BDI | one month
  Change from baseline in the Hospital Anxiety and Depression Scale (HAD), supplemented with a Beck Depression Index (BDI)
BDI | one month
  Change from baseline in the Beck Depression Index (BDI)
CIS | one month
  Change from baseline in the Checklist Individual Strength
TAP | one month
  Change from baseline assessment of alertness and mental flexibility during a Test of Attentional Performance (TAP)
Goal Attainment Scale | one month
  Assessment of pre-defined goal attainment during each treatment period
Registration of Motor Activity and Sleeping pattern | one month
  During each treatment period a continuous registration of Motor Activity and Sleeping pattern by accelerometer, assessing sleep quality, quantity and overall motor activity
Vital Signs | one month
  Change from Baseline assessment of vital signs (heart rate, blood pressure)
ECG | one month
  Change from Baseline assessment of ECG-intervals
Clinical Laboratory | one month
  Change from Baseline assessment of Clinical Laboratory parameters
Pharmacokinetics of KH176 and metabolites | one month
  Attainment of steady state and total exposure (AUC) at steady state conditions
Pharmacokinetics of KH176 and metabolites | one month
  Attainment of steady state and maximal concentrations (Cmax) at steady state conditions
Glutathione | one month
  Change from baseline assessment of the ratio of oxidized/reduced glutathione in blood samples (GSH/GSSG)
Blood biomarker FGF21 | one month
  Change from baseline assessment of FGF21
Blood biomarker GDF15 | one month
  Change from baseline assessment of GDF15
Blood biomarker PRDX1 | one month
  Change from baseline assessment of PRDX1

CONTACTS AND LOCATIONS:
Locations (1):
- Radboud University Medical Center, Nijmegen, Netherlands

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Janssen MCH, Koene S, de Laat P, Hemelaar P, Pickkers P, Spaans E, Beukema R, Beyrath J, Groothuis J, Verhaak C, Smeitink J. The KHENERGY Study: Safety and Efficacy of KH176 in Mitochondrial m.3243A>G Spectrum Disorders. Clin Pharmacol Ther. 2019 Jan;105(1):101-111. doi: 10.1002/cpt.1197. Epub 2018 Sep 3. PMID 30058726